CLINICAL TRIAL: NCT04431466
Title: Phase 2 Clinical Trial to Compare the Efficacy and Safety of Different Doses of Ivermectin in Patients Diagnosed With the New Coronavirus Infection (SARS-CoV-2)
Brief Title: A Study to Compare the Efficacy and Safety of Different Doses of Ivermectin for COVID-19
Acronym: IFORS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Preliminary data from a pilot study suggest that the administration of ivermectin in patients with SARS-CoV-2 is safe, reducing symptoms and viral load. The antiviral effects of ivermectin appear to depend on the dose administered.
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Henrique Pott Junior, Professor, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFORS
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Coronavirus Infection
Keywords: coronavirus infections; SARS-CoV-2; COVID-19; ivermectin; clinical trial
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Ivermectin; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of care (Active Comparator): Standard of care (SOC) treatment
  Interventions: Other: Standard of Care
- SOC plus ivermectin 100 mcg/kg (Experimental): SOC plus ivermectin 100 mcg/kg
  Interventions: Drug: Ivermectin
- SOC plus ivermectin 200 mcg/kg (Experimental): SOC plus ivermectin 200 mcg/kg
  Interventions: Drug: Ivermectin
- SOC plus ivermectin 400 mcg/kg (Experimental): SOC plus ivermectin 400 mcg/kg
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — SOC plus different dosing regimens of Ivermectin
  Arms: SOC plus ivermectin 100 mcg/kg; SOC plus ivermectin 200 mcg/kg; SOC plus ivermectin 400 mcg/kg
Other: Standard of Care — Standard treatment for COVID-19
  Arms: Standard of care

SUMMARY:
In December 2019, a group of patients with pneumonia of unknown cause was linked to a wholesale seafood market in Wuhan, China. The genetic analysis of samples from the lower respiratory tract of these patients indicated a new coronavirus as the causative agent, which was named SARS-CoV-2. The virus spread rapidly to more than 45 countries, including Brazil, causing an international alarm. However, in spite of its epidemiological magnitude, so far, there is no antiviral treatment or vaccine approved for the treatment of this infection. With about 15% to 20% of SARS-CoV-2 patients suffering from serious illnesses and overburdened hospitals, therapeutic options are desperately needed. So, instead of creating compounds from scratch that can take years to develop and test, researchers and public health agencies have sought to redirect drugs already approved for other diseases and known to be widely safe. In this context, the analysis of the international literature shows the existence of an in vitro antiviral activity of ivermectin against SARS-CoV-2. However, there are no studies that have evaluated its clinical effectiveness in patients diagnosed with SARS-CoV-2 infection. Therefore, and considering this knowledge gap, the present study aims to determine the clinical efficacy and safety of different doses of ivermectin in patients diagnosed with SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infection by SARS-CoV-2:

  1. symptoms of acute respiratory tract infection (sudden onset of at least one of the following: cough, fever, shortness of breath) and biomolecular diagnosis of SARS-CoV-2 infection; OR
  2. any acute respiratory disease AND biomolecular diagnosis of SARS-CoV-2 infection; OR
  3. severe acute respiratory infection (fever and at least one sign / symptom of respiratory disease eg cough, fever, shortness of breath) AND in need of hospitalization AND biomolecular diagnosis of SARS-CoV-2 infection;
* Eastern Cooperative Oncology Group Performance Status score 0 to 1;
* National Early Warning Score 0 to 4;
* Ability to understand and consent to participate in this clinical trial, manifested by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* Inability to ingest / absorb the study drug orally through spontaneous ingestion or use of gastro / enteral tubes;
* Any finding of clinical observation (history / physical evaluation) that is interpreted by the investigating physician as a risk to participate in the trial;
* Any laboratory test findings that the investigating physician considers as a risk to the research participant as to his / her participation in the clinical study;
* Any ECG examination finding that the investigating physician considers as a risk to the research participant as to his / her participation in the trial;
* Known hypersensitivity to the components of the drugs used during the study;
* Women in pregnancy or breastfeeding;
* Body weight less than 15kg;
* Estimated glomerular filtration rate (CKD-Epidemiology Collaboration, CKD-EPI) <30 mL / min;
* Aspartate aminotransaminase (AST) or alanine aminotransaminase (ALT)> 5 times the upper limit of normality;
* Refusal to participate;
* Refusal to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Undetectable viral load during 7 days of follow-up. | 7 days following intervention
  Proportion of patients who achieved undetectable viral load during 7 days of follow-up.

SECONDARY OUTCOMES:
Viral load variation in the nasopharyngeal swab. | 7 days following intervention.
  Viral load variation in the nasopharyngeal swab during treatment.
Time to undetectable SARS-CoV-2 viral load in the nasopharyngeal swab. | 7 days following intervention.
  Variation of serum lymphocyte counts during treatment.
Incidence of Treatment-Emergent Self-reported Adverse Events | 28 days following intervention.
  Incidence of Treatment-Emergent Adverse Events as assessed by clinical history and physical examination
Incidence of Treatment-Emergent Laboratory-based Adverse Events | 28 days following intervention.
  Incidence of Treatment-Emergent Adverse Events as assessed by laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Pott Junior, MD PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (2):
- Brazil (2):
  - Hospital Univeristário da Universidade Federal de São Carlos (HU-UFSCar), São Carlos, São Paulo
  - Hospital Universitário da Universidade Federal de São Carlos (HU-UFSCar), São Carlos, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pott-Junior H, Paoliello MMB, Miguel AQC, da Cunha AF, de Melo Freire CC, Neves FF, da Silva de Avo LR, Roscani MG, Dos Santos SS, Chacha SGF. Use of ivermectin in the treatment of Covid-19: A pilot trial. Toxicol Rep. 2021;8:505-510. doi: 10.1016/j.toxrep.2021.03.003. Epub 2021 Mar 9. PMID 33723507 (Retraction: PMID 35528725 Toxicol Rep. 2022 May 02;9:1023)
- See also: Hospital Universitário da UFSCar — http://www2.ebserh.gov.br/web/hu-ufscar